CLINICAL TRIAL: NCT04719741
Title: Drug and Dosage Adjustment in Preventing Postoperative Nausea and Vomiting in Adult Patients Undergoing Elective Surgery Under General Anesthesia
Brief Title: Drug and Dose Adjustment in Preventing Postoperative Nausea and Vomiting
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jordan Hospital (Other)
Responsible Party: Principal Investigator, AbdulRhman MA. M. Ibnouf, Dr., Jordan Hospital
Other Study IDs: JHANES000001
Record Dates: First submitted 2021-01-17; First posted 2021-01-22 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: nausea; vomiting; postoperative; dose adjustment
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (13):
- O-4PI: 4 mg Ondansetron given Pre-Induction
  Interventions: Other: Parallel Assignment
- O-8PI: 8 mg Ondansetron given Pre-Induction
  Interventions: Other: Parallel Assignment
- O-4PE: 4 mg Ondansetron given Pre-Emergence
  Interventions: Other: Parallel Assignment
- O-8PE: 8 mg Ondansetron given Pre-Emergence
  Interventions: Other: Parallel Assignment
- D-4PI: 4 mg Dexamethasone given Pre-Induction
  Interventions: Other: Parallel Assignment
- D-8PI: 8 mg Dexamethasone given Pre-Induction
  Interventions: Other: Parallel Assignment
- D-4PE: 4 mg Dexamethasone given Pre-Emergence
  Interventions: Other: Parallel Assignment
- D-8PE: 8 mg Dexamethasone given Pre-Emergence
  Interventions: Other: Parallel Assignment
- O-4PI+D-8PI: 4 mg Ondansetron pre-induction+ 8 mg Dexamethasone pre-induction
  Interventions: Other: Parallel Assignment
- O-4PI+D-8PE: 4 mg Ondansetron pre-induction+ 8 mg Dexamethasone pre-emergence
  Interventions: Other: Parallel Assignment
- O-4PE+D-8PI: 4 mg Ondansetron pre-emergence + 8 mg Dexamethasone pre-induction
  Interventions: Other: Parallel Assignment
- O-4PE+D-8PE: 4 mg Ondansetron pre-emergence + 8 mg Dexamethasone pre-emergence
  Interventions: Other: Parallel Assignment
- Placebo Group: 2 ml Saline 0.9%
  Interventions: Other: Parallel Assignment

INTERVENTIONS:
Other: Parallel Assignment — Prospective, Triple blinded, randomized, controlled trial

SUMMARY:
The aim is to evaluate the effectiveness of different regimens of prophylactic Ondansetron, Dexamethasone, or both, on the incidence and severity of post-operative nausea and vomiting.

DETAILED DESCRIPTION:
Patients will be randomized to one of four arms: Ondansetron (4O-PE: 4 mg Ondansetron pre-emergence, 8O-PE: 8 mg Ondansetron pre-emergence, 4O-PI: 4 mg Ondansetron pre-incision, 8O-PI: 8 mg Ondansetron pre-incision), Dexamethasone (4D-PE: 4 mg Dexamethasone pre-emergence, 8D-PE: 8 mg Dexamethasone pre-emergence, or 4D-PI: 4 mg Dexamethasone pre-incision, or 8D-PI: 8 mg Dexamethasone pre-incision), Combination Therapy group (4O-PI+8D-PI: 4 mg Ondansetron pre-incision + 8 mg Dexamethasone pre-incision, 4O-PI+8D-PE: 4 mg Ondansetron pre-incision + 8 mg Dexamethasone pre-emergence, 4 O-PE+8D-PI: 4 mg Ondansetron pre-emergence + 8 mg Dexamethasone pre-induction, 4 O-PE+8D-PE: 4 mg Ondansetron pre-emergence + 8 mg Dexamethasone pre-emergence), and Placebo group 2 ml Saline 0.9%. Primary outcome will be the incidence of PONV in the PACU prior to discharge.

ELIGIBILITY:
Inclusion Criteria:

* ASA grade I and II
* Aged 18-70 years
* Patients scheduled for elective surgery under general anesthesia

Exclusion Criteria:

* All patients who received antiemetics or cortisone within 48 hr before surgery
* Pregnant, breast feeding ladies
* Any patient with BMI (Body Mass Index) > 34 kg/m²
* Patient with gastrointestinal, hepatic, renal, mental or psychiatric illnesses were also excluded from the study protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-05-20 (Estimated); Study Completion 2024-08-20 (Estimated)

PRIMARY OUTCOMES:
Presence of postoperative nausea and/or vomiting | 24 hours
  Follow if the patient complained about postoperative nausea and/or vomiting in terms of use of antiemetic drugs

CONTACTS AND LOCATIONS:
Overall Officials: AbdulRhman MA Ibnouf, MBBS, Study Director — Anaesthesia Department, Jordan Hospital
Locations (1):
- Jordan Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided